CLINICAL TRIAL: NCT06721338
Title: Safety and Efficacy of Mechanical Thrombectomy Utilizing Reversal Flow
Brief Title: Mechanical Thrombectomy Blood Flow Reversal
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to resume the study due to patient billing issues. No actual clinical reason.
Sponsor: MediSys Health Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2245475
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Large Vessel Occlusion
Keywords: stroke; large vessel occlusion; blood flow reversal; mechanical thrombectomy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Stroke patients with LVO (Experimental): Eligible patients for the study will be stroke patients with large vessel occlusion who meet inclusion criteria.
  * Age > 18-year-old
  * Last known well less than 24 hours
  * Large vessel occlusion of intra-cranial ICA or MCA M1 segment
  * ASPECTS of 4 or above
  * Baseline modified Rankin scale of 3 or less.
  * More than 20 ml penumbra on CTP
  * Less than 100 ml infarct core on CTP
  Before the mechanical thrombectomy is completed, a surgical cut will be made to the other groin that has not been operated on. A catheter and wire are used to access the newly punctured femoral vein. A device called an aspiration filter will connect a catheter from your femoral vein to an aspiration catheter at the target site. Once this connection is complete, full removal of the blockage by the stent retriever will occur while blood flow is reversed.
  Interventions: Device: Mechanical thrombectomy via blood flow reversal using BOBBY balloon guide catheter

INTERVENTIONS:
Device: Mechanical thrombectomy via blood flow reversal using BOBBY balloon guide catheter — After 2 min. of mechanical thrombectomy (MT), the side port of a BOBBY balloon guide catheter will be flushed again with heparin and the balloon deflated. A follow up angiogram will be performed to determine whether to proceed with another MT pass using the same procedure or to stop if successful recanalization has been achieved. At the end of the procedure, multiple angiograms will be performed and used to record the final TICI score. Angiograms of neck vessels will be used to rule out complications. Groin angiograms will evaluate the puncture site before closure. The catheters will then be removed, allowing hemostasis to be achieved in the groin. An angioseal closure device will be used on the arterial site if not contraindicated and a venous Vascade for the venous side.

SUMMARY:
The goal of this study is to reduce the chance of complications during mechanical thrombectomy, which is a procedure to remove blockages from the brain. This study is combining two established and standard procedures for the first time so that the patient may benefit from both and reduce the chance of another stroke during the procedure. Our main goal is to show that this combination is safe, feasible, and effective for stroke patients.

The combined procedures are described as follows:

1. Mechanical Thrombectomy: while the patient is asleep under light or general anesthesia, a surgical cut will be made in their groin to access the common femoral artery. A catheter will be inserted into this cut so that a wire can advance through the artery. Using an imaging technique called angiography, a blueprint is used to advance the wire from an artery in their groin, to their neck, into their brain and locate the target blockage. Once the target is located, more wires and catheters are used to finetune the extraction process. A stent retriever is placed on standby before removing the blockage.
2. Reversal Flow: before the mechanical thrombectomy is completed, a surgical cut will be made to the other groin that has not been operated on. A catheter and wire are used to access the newly punctured femoral vein. A device called an aspiration filter will connect a catheter from their femoral vein to an aspiration catheter at the target site. Once this connection is complete, full removal of the blockage by the stent retriever will occur while blood flow is reversed.

DETAILED DESCRIPTION:
BACKGROUND Stroke is an acute injury to the brain with a vascular cause that results in permanent neuronal injury and functional disability. Stroke can be divided into two subtypes: ischemic and hemorrhagic. Ischemic strokes occur when an occlusion (i.e., blockage of blood vessel) or flow-limiting stenosis of cerebral vessels (i.e., narrowing of an artery in the brain) cause inadequate blood flow for neuronal sustainment. They are caused by cerebral small vessel disease, cardioembolism, and large artery disease. Hemorrhagic strokes typically result from a rupture caused by an aneurysm or other non-traumatic causes (e.g., chronic hypertension) and from illicit drug abuse.

Globally, stroke is the second leading cause of both death and disability. In 2016, worldwide prevalence was 80.1 million, and slightly higher among women (41.1 million) than in men (39.0 million). The incidence of new strokes globally in 2016 was 13.7 million. In the United States, stroke is the fifth-leading cause of death and a major cause of severe disability, as well as the primary cause of hospitalization for neurologic disease. Within the US, the prevalence of stroke is approximately 3% in adults 20 years or older, translating to approximately 7 million occurrences of stroke within this population. Of all strokes, approximately 87% are ischemic. In 2017, the global incidence of ischemic strokes was 101.3 per 100,000 people.

Certain factors, both modifiable and non-modifiable, can increase an individual's likelihood of stroke. The most prominent non-modifiable risk factor is age. Incidence doubles for each decade after the age of 55, increasing the risk for individuals within this age group. Other key non-modifiable risk factors include sex, ethnicity, and genetics. The most important modifiable risk factor for stroke is hypertension. Elevated blood pressure increases the risk of stroke; half of all stroke patients have a history of hypertension. Other notable modifiable risk factors include diabetes mellitus, cardiac factors (e.g., atrial fibrillation), smoking, high alcohol consumption, substance abuse, obesity, and inflammation.

Stroke can have a monumental effect on many areas of life, both individually and globally. Stroke survivors develop physical impairments which can limit daily living, as well as communication skills. Additionally, approximately 80% of the stroke population experience cognitive impairments, which has a sizeable effect on an individual's ability to complete daily tasks. Physical consequences of stroke can impede survivors from participating in work or other activities that were at one point an essential part of their identity. Aside from physical effects, stroke can also greatly impact one's mental state. Additionally, variations in communication skills caused by stroke have a profound effect on self-confidence. As a result, stroke survivors engage in less social activities, causing a substantial vulnerability to their social networks. Furthermore, the economic burden associated with stroke is vast, with the 2019 global value of lost welfare due to stroke being $2059.67 billion. Addressing stroke care and developing new targeted approaches to aid in stroke treatment can have a lasting benefit not only to the individual, but also worldwide.

Reperfusion therapy can be used to treat ischemic stroke, as it allows for the restoration of blood flow to salvageable brain tissue. Reperfusion therapy has two main components: thrombolysis, including intravenous (IV) tissue plasminogen activator (tPA), and endovascular interventions such as mechanical thrombectomy. The two components of reperfusion therapy, thrombolysis and endovascular interventions, can be used separately or in tandem. Thrombolysis is a pharmacological treatment to dissolve blood clots using an infusion of tPA, known as alteplase. The only FDA-approved IV thrombolytic agent for the treatment of an ischemic stroke is alteplase, yet off-label IV tenecteplase, a genetically modified form of alteplase given as a single bolus, is beginning to be used more regularly. Some guidelines have recommended either alteplase or tenecteplase for patients with acute ischemic stroke within 4.5 hours after known onset. It is crucial to deliver IV thrombolysis expeditiously, as the number needed to treat for favorable outcome almost double from 5 (for treatment within 90 min) to 9 (when given at 3-4.5 hours). However, the benefits of IV tPA varies among those with severe stroke caused by large artery occlusion due to an inability to achieve early recanalization (i.e., restoration of blood flow). Significant independent risk factors predicting poor outcomes post IV-thrombolysis are length and location of the arterial thrombus (i.e., blood clot). Therefore, this lack of efficacy of what was once the only treatment for stroke led to efforts to remove larger arterial thrombi using intra-arterial techniques by mechanical thrombectomy, the other component of reperfusion therapy.

A paradigm shift in treatment of acute ischemic stroke in recent years favoring endovascular reperfusion technique is due to the results of many positive trials. One such trial, MR CLEAN, showed a significant absolute benefit of mechanical thrombectomy in patients with large vessel occlusion (LVO). Soon after, subsequent trials such as ESCAPE, SWIFT PRIME, REVASCAT, THRACE, and PISTE were conducted and concluded the same. Thus, the American Stroke Association amended the 2013 guidelines in 2015 to include mechanical thrombectomy as the standard of care in patients with LVO presenting within 6 hours of last known well or symptom initiation. In 2018, the guidelines endorsed inclusion of the delayed window period treatment for endovascular reperfusion, which states that IV thrombolysis is only given with 3-4.5 hours after known onset, while mechanical thrombectomy can be done up to 72 hours after last known well.

The "time is brain" edict (i.e., time is of the essence when treating a stroke) holds true for mechanical thrombectomy, in that early reperfusion and the extent of reperfusion affect the outcome in LVO. The techniques involve deployment of a stent retriever (i.e., metal stent that grabs and extracts blood clots in blocked arteries), a large-bore catheter for distal aspiration (i.e., tube used to draw out a blockage further away), or a combination of the two with or without a balloon guide catheter (BGC). BGCs can be beneficial during clot retrieval by creating proximal blood flow arrest, reducing embolic burden (blockage in blood vessel causing embolism), and shortening procedure time. The standard technique is conducted by first placing the guide catheter in the internal carotid artery (ICA), then using a microcatheter to advance over a microwire through an aspiration catheter and cross the occlusion by passing through the thrombus. The microwire is then withdrawn, and a contrast injection is performed to evaluate the distal arterial segment and confirm the tip of the microcatheter is distal to the thrombus. A stent retriever is then advanced in the microcatheter and deployed across the thrombus by gradually unsheathing the microcatheter. This allows for immediate flow restoration in the previously occluded vascular territory. Then, aspiration starts through the aspiration catheter to help with engaging the clot. After a few minutes of thrombus integration in the stent retriever, the stent retriever is then slowly and carefully withdrawn into the guide/aspiration catheter and removed. While crossing the clot with catheters or while removing it from the brain vessels, there is a chance of dislodging some part of the clot, causing distal embolization, which would worsen the patient's outcome and increase stroke burden.

One of the main proposed etiologies for distal embolism is the anterograde blood flow around the aspiration catheter that may send fragments of the clot distally. Using larger aspiration catheters and inflating BGCs to achieve flow arrest have reduced the chances of distal emboli, but not completely. The main explanation for this is that despite arresting or reducing the blood flow, there would still be "anterograde" circulation through the intra-cranial arteries from collateral circulations, such as through anterior or posterior communicating arteries. However, there are currently established techniques to reverse intra-cranial blood circulation during extra-cranial internal carotid artery stenting. The Trans-Carotid Arterial Revascularization (TCAR) procedure applies blood flow reversal from the carotid artery to the contralateral femoral vein through a filter while deploying the stent in ICA. This flow reversal has been shown to be effective in reducing the chance of distal emboli and silent stroke from 40% to 17%. Our proposed technique in this study is to combine blood flow reversal, like the TCAR procedure, with standard thrombectomy to reduce the chance of distal embolism and improve the patient's outcome. Our technique will include a BGC, which is positioned in the ICA. The BGC is inflated to achieve flow arrest and prevent thrombus dislodgement and distal embolization during removal of the stent retriever.

Mechanical thrombectomy alone reduces disability in LVO patients (adjusted odds ratio [OR]: 2.49) and the number needed to treat for a reduction of disability by at least one point on the modified Rankin scale is 2.6. Many trials, such as MR CLEAN, DAWN, and DEFUSE3, found a substantial increase in lifetime quality-adjusted life years using mechanical thrombectomy. Despite their clear benefits, these standard procedures still carry the risk of distal emboli formation, which can worsen stroke outcomes. About two in every five cases experience distal emboli, which produces lower rates of complete reperfusion, larger final infarct volumes, and worse functional outcomes. The proposed technique aims to improve the efficacy of performing mechanical thrombectomy utilizing a reverse flow technique with the hope of reducing distal emboli and improving first-pass success rate compared with standard technique. As the first phase of trial, this study is designed to prove feasibility and safety of flow reversal thrombectomy. This study will show a separate way to utilize approved mechanical thrombectomy procedures so that they will be more effective, improving favorable outcomes for this acute stroke treatment.

PROCEDURES

OVERVIEW:

The goal of this study is to evaluate the safety and feasibility of endovascular mechanical thrombectomy under "blood flow reversal". To accomplish this goal, 20 patients from Jamaica Hospital Medical Center (JHMC) undergoing mechanical thrombectomy would be enrolled in our study and the safety of the procedure will be evaluated. Patients would be followed for approximately 3 months post-procedure.

The study is an event specific procedure. Patients presenting with clinical symptoms of stroke (e.g., weakness, aphasia, facial droop, gaze deviation, altered mental status, etc.) within 24 hours of the time when the patient was last seen without stroke symptoms or at their baseline health (based on the report of the patient, witness, or family members), will be assessed for mechanical thrombectomy eligibility.

This assessment will be conducted by the neurointerventional proceduralist using the study's inclusion and exclusion criteria. Once a patient meets eligibility criteria, the neurointerventionalist (NI) will discuss the purpose of the study and how the reverse flow procedure is modified from standard of care, its risks and benefits, and the transition of care after the conclusion of the procedure with the patient or family either via phone or in-person according to the consent form. After this conversation, the NI will obtain either assent or consent. The patient will then be transported to the intervention laboratory as per hospital protocol.

At the intervention laboratory, the procedure will be performed under conscious sedation or generalized anesthesia based on the patient's condition (i.e., underlying comorbidity, mental status, complexity of the procedure) and discussions between the anesthesiologist and NI. Pulse oximetry will be monitored by placing a pulse oximeter on both lower extremities (toes). Distal pulses will be checked manually and with a Doppler ultrasound.

An 8-Fr Destination 45 cm sheath (Terumo, Japan) will be used for arterial access of the right or left common femoral artery. Then, a Bobby balloon guide catheter 95 cm (Terumo Neuro, USA) will advance over a select catheter and over a 038 Terumo glidewire (Terumo, Japan) to allow the left or right common carotid artery to be selected. After the baseline angiography, the guide catheter will be advanced into the high cervical ICA under roadmap, which is a processed angiography image showing brain vessels under which interventionist could navigate catheters and wires. Baseline angiogram will be performed based on which appropriate aspiration (6-Fr or 5-Fr Sofia, Terumo Neuro) and microcatheter (Headway 27, Terumo Neuro) are selected and advanced over the 014-024 microguidewire intra-cranially, as well as whether the embolus is engaged with aspiration with or without stent retriever deployment.

Then, an aspiration catheter will be left in place for 3-5 minutes. At this time, the contralateral femoral vein will be punctured, and a 6-Fr short sheath (Terumo, Japan) will be inserted. The side port of the guide catheter will be connected through an aspiration filter (Imperative Care, USA) to the venous sheath. Before retrieving the aspiration catheter, the guide catheter balloon will be inflated to achieve flow arrest, and its side port will be opened to the venous side to achieve flow reversal. The aspiration catheter will then be removed in standard fashion to complete the thrombectomy pass. Then, flow reversal will be allowed for 2 minutes.

After two minutes, the side port of the guide catheter will be placed on heparinized flush again and the balloon will be deflated. A follow up angiogram will be performed, which will determine whether to proceed with another thrombectomy pass following the same procedure or to halt the procedure if successful recanalization has been achieved. At the conclusion of the procedure, multiple angiograms will be performed. The final angiograms in standard anterior-posterior (AP) and lateral will be used to record the final TICI score. Angiograms of neck vessels will be obtained to rule out complications, such as dissection or vasospasm. Groin angiograms will be performed to evaluate the puncture site before using the closure device. The catheters will then be removed, allowing hemostasis to be achieved in the groin. An angioseal closure device will be used on the arterial site if not contra-indicated and a venous Vascade closure device will be used for the venous side.

The procedure's duration will depend on the patient's cerebrovascular anatomy, comorbid conditions, and the clot's nature, but is approximately 30 minutes. The goal of our modified procedure is the absence of distal emboli post procedure and a reperfusion with a modified Thrombolysis in Cerebral Infarction (mTICI) score of ≥2b. A TICI Score is a tool used to grade how well the blood flow was restored in your brain's circulation after the blood clot was removed. The score ranges from 0 to 3, but the acceptable score is ≥2b.

Procedural complications, venous puncture related complications, procedure outcome, post op NIHSS, discharge NIHSS, post-op brain MRI, doppler of lower extremities, length of hospital stay, and disposition would be recorded. The patient will be followed up after the procedure, and a follow up appointment at 30 and 90 days after discharge. During follow-up visits in the Stroke Clinic, a general neuroassessment will be performed, along with National Institute of Health Stroke Scale (NIHSS) and Modified Rankin Scale (mRS).

TIMELINE:

This procedure is a modification of the standard practice to limit the complication of distal emboli. As an acute treatment for acute ischemic stroke, the length of the procedure will vary, depending on patient's cerebrovascular anatomy, comorbidity, and stroke severity but, on average is less than 30 minutes from skin puncture. The patient will then be cared for in the intensive care unit for close monitoring, then transferred to stroke unit after 24 hours, provided that neurological status and vital signs are within parameters. During hospitalization, the patient will be worked up to look for stroke etiology. Once the workup is done, the patient will be discharged based on the recommendation of the physiatrist or neurologist.

Post-discharge, the patient will have a 30-day, 90-day, and 3 months follow up appointments, which will be scheduled prior to discharge. The sessions will be at least 20-30 minutes, where the patient will be assessed for current neurological and functional status. A modified Rankin Scale (mRS) and National Institute of Health Stroke Scale (NIHSS) scores will be obtained and documented.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18-year-old
* Last known well less than 24 hours
* Large vessel occlusion of intra-cranial ICA or MCA M1 segment
* ASPECTS of 4 or above
* Baseline modified Rankin scale of 3 or less.
* More than 20 ml penumbra on CTP
* Less than 100 ml infarct core on CTP

Exclusion Criteria:

• Large vessel occlusion on the posterior circulation, with tandem occlusion, has known history of patent foramen ovale, has deep venous thrombosis of lower extremity, absent family members to consent, large established stroke on CT/CT Perfusion with ASPECTS <5, the individual consenting is a non-English speaker, and poor baseline function will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of Treatment Defined by the Abscence of Distal Emboli and a mTICI score of ≥2b per Participant Post-Procedure | From enrollment to the end of treatment at 3 months
  Whether this experimental procedure (blood flow reversal) on performing acute intervention (mechanical thrombectomy) for stroke is feasible, measured by the absence of distal emboli post procedure (measured as a continuous variable with none being 0) and a reperfusion with a modified Thrombolysis in Cerebral Infarction (mTICI) score of ≥2b. A TICI Score is a tool used to grade how well the blood flow was restored in the brain's circulation after the blood clot was removed. The score ranges from 0 to 3, but the acceptable score is ≥2b.

CONTACTS AND LOCATIONS:
Locations (1):
- Jamaica Hospital Medical Center, Jamaica, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saver JL, Chaisinanunkul N, Campbell BCV, Grotta JC, Hill MD, Khatri P, Landen J, Lansberg MG, Venkatasubramanian C, Albers GW; XIth Stroke Treatment Academic Industry Roundtable. Standardized Nomenclature for Modified Rankin Scale Global Disability Outcomes: Consensus Recommendations From Stroke Therapy Academic Industry Roundtable XI. Stroke. 2021 Aug;52(9):3054-3062. doi: 10.1161/STROKEAHA.121.034480. Epub 2021 Jul 29. PMID 34320814
- [Background] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Background] Sarre S, Redlich C, Tinker A, Sadler E, Bhalla A, McKevitt C. A systematic review of qualitative studies on adjusting after stroke: lessons for the study of resilience. Disabil Rehabil. 2014;36(9):716-26. doi: 10.3109/09638288.2013.814724. Epub 2013 Jul 25. PMID 23883420
- [Background] Saini V, Guada L, Yavagal DR. Global Epidemiology of Stroke and Access to Acute Ischemic Stroke Interventions. Neurology. 2021 Nov 16;97(20 Suppl 2):S6-S16. doi: 10.1212/WNL.0000000000012781. PMID 34785599
- [Background] Saa JP, Tse T, Baum C, Cumming T, Josman N, Rose M, Carey L. Longitudinal evaluation of cognition after stroke - A systematic scoping review. PLoS One. 2019 Aug 29;14(8):e0221735. doi: 10.1371/journal.pone.0221735. eCollection 2019. PMID 31465492
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Parthasarathy R, Gupta V. Mechanical Thrombectomy: Answering Unanswered. Ann Indian Acad Neurol. 2020 Jan-Feb;23(1):13-19. doi: 10.4103/aian.AIAN_359_19. PMID 32055116
- [Background] Northcott S, Moss B, Harrison K, Hilari K. A systematic review of the impact of stroke on social support and social networks: associated factors and patterns of change. Clin Rehabil. 2016 Aug;30(8):811-31. doi: 10.1177/0269215515602136. Epub 2015 Sep 1. PMID 26330297
- [Background] Murphy SJ, Werring DJ. Stroke: causes and clinical features. Medicine (Abingdon). 2020 Sep;48(9):561-566. doi: 10.1016/j.mpmed.2020.06.002. Epub 2020 Aug 6. PMID 32837228
- [Background] Muir KW, Ford GA, Messow CM, Ford I, Murray A, Clifton A, Brown MM, Madigan J, Lenthall R, Robertson F, Dixit A, Cloud GC, Wardlaw J, Freeman J, White P; PISTE Investigators. Endovascular therapy for acute ischaemic stroke: the Pragmatic Ischaemic Stroke Thrombectomy Evaluation (PISTE) randomised, controlled trial. J Neurol Neurosurg Psychiatry. 2017 Jan;88(1):38-44. doi: 10.1136/jnnp-2016-314117. Epub 2016 Oct 18. PMID 27756804
- [Background] Mishra SM, Dykeman J, Sajobi TT, Trivedi A, Almekhlafi M, Sohn SI, Bal S, Qazi E, Calleja A, Eesa M, Goyal M, Demchuk AM, Menon BK. Early reperfusion rates with IV tPA are determined by CTA clot characteristics. AJNR Am J Neuroradiol. 2014 Dec;35(12):2265-72. doi: 10.3174/ajnr.A4048. Epub 2014 Jul 24. PMID 25059699
- [Background] Luk Y, Chan YC, Cheng SW. Transcarotid Artery Revascularization as a New Modality of Treatment for Carotid Stenosis. Ann Vasc Surg. 2020 Apr;64:397-404. doi: 10.1016/j.avsg.2019.11.001. Epub 2019 Nov 6. PMID 31705988
- [Background] Li S, Gu HQ, Li H, Wang X, Jin A, Guo S, Lu G, Che F, Wang W, Wei Y, Wang Y, Li Z, Meng X, Zhao X, Liu L, Wang Y; RAISE Investigators. Reteplase versus Alteplase for Acute Ischemic Stroke. N Engl J Med. 2024 Jun 27;390(24):2264-2273. doi: 10.1056/NEJMoa2400314. Epub 2024 Jun 14. PMID 38884332
- [Background] Kim SH, Choi JH, Kang MJ, Cha JK, Kim DH, Nah HW, Park HS, Kim SH, Huh JT. Efficacy of Combining Proximal Balloon Guiding Catheter and Distal Access Catheter in Thrombectomy with Stent Retriever for Anterior Circulation Ischemic Stroke. J Korean Neurosurg Soc. 2019 Jul;62(4):405-413. doi: 10.3340/jkns.2019.0007. Epub 2019 Jul 1. PMID 31290296
- [Background] Katsanos AH, Psychogios K, Turc G, Sacco S, de Sousa DA, De Marchis GM, Palaiodimou L, Filippou DK, Ahmed N, Sarraj A, Menon BK, Tsivgoulis G. Off-Label Use of Tenecteplase for the Treatment of Acute Ischemic Stroke: A Systematic Review and Meta-analysis. JAMA Netw Open. 2022 Mar 1;5(3):e224506. doi: 10.1001/jamanetworkopen.2022.4506. PMID 35357458
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Hirano T, Sasaki M, Mori E, Minematsu K, Nakagawara J, Yamaguchi T; Japan Alteplase Clinical Trial II Group. Residual vessel length on magnetic resonance angiography identifies poor responders to alteplase in acute middle cerebral artery occlusion patients: exploratory analysis of the Japan Alteplase Clinical Trial II. Stroke. 2010 Dec;41(12):2828-33. doi: 10.1161/STROKEAHA.110.594333. Epub 2010 Oct 28. PMID 21030700
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Gerstl JVE, Blitz SE, Qu QR, Yearley AG, Lassaren P, Lindberg R, Gupta S, Kappel AD, Vicenty-Padilla JC, Gaude E, Atchaneeyasakul KC, Desai SM, Yavagal DR, Peruzzotti-Jametti L, Patel NJ, Aziz-Sultan MA, Du R, Smith TR, Bernstock JD. Global, Regional, and National Economic Consequences of Stroke. Stroke. 2023 Sep;54(9):2380-2389. doi: 10.1161/STROKEAHA.123.043131. Epub 2023 Jul 27. PMID 37497672
- [Background] Feske SK. Ischemic Stroke. Am J Med. 2021 Dec;134(12):1457-1464. doi: 10.1016/j.amjmed.2021.07.027. Epub 2021 Aug 27. PMID 34454905
- [Background] Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, Brott T, Cohen G, Davis S, Donnan G, Grotta J, Howard G, Kaste M, Koga M, von Kummer R, Lansberg M, Lindley RI, Murray G, Olivot JM, Parsons M, Tilley B, Toni D, Toyoda K, Wahlgren N, Wardlaw J, Whiteley W, del Zoppo GJ, Baigent C, Sandercock P, Hacke W; Stroke Thrombolysis Trialists' Collaborative Group. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a meta-analysis of individual patient data from randomised trials. Lancet. 2014 Nov 29;384(9958):1929-35. doi: 10.1016/S0140-6736(14)60584-5. Epub 2014 Aug 5. PMID 25106063
- [Background] Chueh JY, Kang DH, Kim BM, Gounis MJ. Role of Balloon Guide Catheter in Modern Endovascular Thrombectomy. J Korean Neurosurg Soc. 2020 Jan;63(1):14-25. doi: 10.3340/jkns.2019.0114. Epub 2019 Oct 8. PMID 31591997
- [Background] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Background] Bhatia R, Hill MD, Shobha N, Menon B, Bal S, Kochar P, Watson T, Goyal M, Demchuk AM. Low rates of acute recanalization with intravenous recombinant tissue plasminogen activator in ischemic stroke: real-world experience and a call for action. Stroke. 2010 Oct;41(10):2254-8. doi: 10.1161/STROKEAHA.110.592535. Epub 2010 Sep 9. PMID 20829513
- [Background] Bagley JH, Priest R. Carotid Revascularization: Current Practice and Future Directions. Semin Intervent Radiol. 2020 Jun;37(2):132-139. doi: 10.1055/s-0040-1709154. Epub 2020 May 14. PMID 32419725
- [Background] Bhaskar S, Stanwell P, Cordato D, Attia J, Levi C. Reperfusion therapy in acute ischemic stroke: dawn of a new era? BMC Neurol. 2018 Jan 16;18(1):8. doi: 10.1186/s12883-017-1007-y. PMID 29338750